CLINICAL TRIAL: NCT06204510
Title: Effects of Complex Decongestive Therapy on Proprioception, Balance and Tactile Sense in Lymphedema After Cancer Surgery: A Prospective Randomized Controlled Study
Brief Title: Effects of Complex Decongestive Therapy on Proprioception, Balance and Tactile Sense
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Assistant Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/03.01
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Lymphedema of Leg; Sensitisation; Balanced; Therapy-Associated Cancer
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- study group (Experimental)
  Interventions: Other: complex decongestive therapy

INTERVENTIONS:
Other: complex decongestive therapy — This application consists of manual lymph drainage, skin care, compression bandage and exercises. This phase will continue for 3 weeks, 5 days a week.
  Arms: study group

SUMMARY:
The aim of this study is to investigate the effects of complex decongestive physiotherapy (CDP) on propriseception, balance and sensation in patients with secondary lymphedema that develops in the lower extremities after cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having unilateral lymphedema in the lower extremity secondary to cancer surgery

Exclusion Criteria:

* Having bilateral lower extremity lymphedema
* Having an active infection
* Having a mental cognitive disorder
* Being at a level where communication and cooperation cannot be established
* Situations where manual lymphatic drainage is contraindicated (such as severe heart failure and/or uncontrolled rhythm disorder, uncontrolled hypertension, pregnancy, presence of thrombus, active infection)
* Presence of metastasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Proprioception | 10 minutes
  Joint position sense: While the patient lies in the prone position, 15-45-60 degrees of knee flexion will be evaluated in 2 different ways: eyes open and eyes closed. Participants will be asked to find the target angle they have been taught with their eyes closed and will be asked to say "here" in the position where they think they have reached the target angle.
One-leg Standing Test | 5 minutes
  It is performed with one leg supported to evaluate static balance. The eyes will be fixed in the direction of the head and the participant will be asked to close their eyes and will be expected to maintain balance for 30 seconds. It ends when the balance is disrupted. The test will be terminated when the maximum time of 30 seconds expires.
30 Seconds Sit-Stand-on-Chair Test: | 5 minutes
  In the application of the test, the participant will be asked to sit in the middle part of a 43.18 cm (12 inches) high chair with his back upright, his feet on the ground and his arms crossed in front of his body. While in this position, the test started with the "start" command and the participant will be asked to stand up and sit down as fully as he can for 30 seconds. Standing upright once will count as 1, and the number of times he stands upright during 30 seconds will constitute the participant's score
Softt Touch Sense | 5 minutes
  It is evaluated with Semmes Weinstein Monofilaments (SWM). The test will be performed with the patient lying in the supine position. In practice, the areas to be tested will be determined as the 1st metatarsal and 5th metatarsal heads and the midpoint of the heel. Values between 1.65-2.83 (green) are considered normal sensation. Values between 3.22-3.61 (blue) are reduced light touch, values between 3.84-4.31 (purple) are reduced protective sensation, values between 4.56-6.65 (red) are loss of protective sensation and 6, If there is no response to 65, it is considered deep pressure perception.
Two Point Discrimination | 5 minutes
  Participants will be evaluated in a sitting position with eyes closed using an aesthesiometer (Instrument Company, Lafayette, IN, USA). The evaluation will be made from the trans-metatarsal area, the middle of the foot and the middle of the heel. It will start from the range where the two points can be easily distinguished. The shortest length felt between two points will give the static two-point discrimination value.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cihan E, Pirincci CS. The efficacy of complex decongestive therapy in the treatment of lymphedema associated with endometrial and cervical cancer: evaluation of sensation and balance. Support Care Cancer. 2026 Jan 22;34(2):113. doi: 10.1007/s00520-026-10330-9. PMID 41569453